CLINICAL TRIAL: NCT03037710
Title: Link-HF: Multisensor Non-invasive Telemonitoring System for Prediction of Heart Failure Exacerbation
Acronym: LINK-HF
Status: Completed | Type: Observational
Sponsor: Josef Stehlik (Other)
Responsible Party: Sponsor-Investigator, Josef Stehlik, Principal Investigator, University of Utah
Organization: University of Utah (Other)
Other Study IDs: 81833
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Cardiac Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: HealthPatch — A multi-sensor device to collect continuous vital signs

SUMMARY:
This is a multi-center, non-randomized, non-interventional study to evaluate the accuracy of a remote monitoring and analytical platform for prediction of heart failure exacerbation. The platform acquires continuous multivariate vital signs from HF patients using a new ambulatory wearable (attached by an adhesive) multi-sensor device and analyzes the data using a novel machine learning algorithm.

DETAILED DESCRIPTION:
The analytics being investigated includes a Similarity-Based Modeling technique, that empirically estimates the expected physiological behavior of a subject based on prior learned dynamic data, for comparison to actual measured behavior from the subject, to reveal discrepancies hidden by normal variation. The measurements are typically an ensemble of vital signs that effectively characterizes the physiological "control system" of the subject. This technique is multivariate: multiple variables are leveraged, because single variables in isolation have little context - a high heart rate by itself could mean a person is exerting himself, or it could mean his physiology is in distress even though he is not exerting himself. With reference to several other variables, however, such as respiration rate, oximetry and motion/activity, a high heart rate might be recognized as a normal state when accompanied by the corroborating data showing a high respiration rate, a normal oximetry and a high level of motion - the person is exercising.

A wearable adhesive multi-sensor device will be used to collect continuous vital sign and other data from study subjects, including heart rate, respiration rate, bodily motion/activity, skin temperature, pulse, electrocardiogram and peripheral capillary oxygen saturation. Subjects are provided with a smartphone or cellular tablet that will be paired with the multi-sensor device to receive data and upload it to the analytics server via cellular network or WiFi internet. Study staff will interact with the subject during visits scheduled for routine heart failure follow-up to capture pre-specified heart failure medical events. All standard of care clinic and hospitalization notes and procedure reports including echocardiograms, right heart catheterizations, pulmonary function tests, six minute walk tests and radiology reports will be collected as they occur.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 years old or older
2. NYHA( New York Heart Association Functional Classification) Class II-IV, documented in site's medical record system.
3. Subject able and willing to sign Informed Consent Document.
4. Subject willing and able to perform all study related procedures.

Exclusion Criteria:

1. Expected LVAD (Left Ventricular Assist Device) implantation or heart transplantation in the next 30 days.
2. Skin damage or significant arthritis, preventing wearing of device.
3. Uncontrolled seizures or other neurological disorders leading to excessive abnormal movements or tremors in the upper body.
4. Pregnant women or those who are currently nursing.
5. Visual/cognitive impairment that as judged by the investigator does not allow the subject to independently follow rules and procedures of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with heart failure, NYHA Class II-IV
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01-26 (Actual); Study Completion 2017-01-26 (Actual)

PRIMARY OUTCOMES:
Detection of Heart Failure Exacerbation Event | 90 Days
  Correlation of algorithmic alerts generated by a non-invasive telemonitoring system to a verified heart failure exacerbation event, measured in percent accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Josef Stehlik, MD, Principal Investigator — University of Utah
Locations (4):
- United States (4):
  - Palo Alto VA Health Care System, Palo Alto, California
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - George E Wahlen Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stehlik J, Schmalfuss C, Bozkurt B, Nativi-Nicolau J, Wohlfahrt P, Wegerich S, Rose K, Ray R, Schofield R, Deswal A, Sekaric J, Anand S, Richards D, Hanson H, Pipke M, Pham M. Continuous Wearable Monitoring Analytics Predict Heart Failure Hospitalization: The LINK-HF Multicenter Study. Circ Heart Fail. 2020 Mar;13(3):e006513. doi: 10.1161/CIRCHEARTFAILURE.119.006513. Epub 2020 Feb 25. PMID 32093506